CLINICAL TRIAL: NCT02471664
Title: The Study on Safety and Feasibility of Mitral Loop Cerclage(MLC) Annuloplasty Procedure With Investigational Medical Device (MLC-B-45-75-R and Other 11 Models) : Single-centre, Open Label, Single Arm, Feasibility Test
Brief Title: Mitral Loop Cerclage(MLC) for Reducing Functional Mitral Regurgitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tau-MEDICAL Co., Ltd. (Industry)
Responsible Party: Principal Investigator, June-Hong Kim, MD, PhD, Professor, Pusan National University Yangsan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPMMLC
Record Dates: First submitted 2015-06-05; First posted 2015-06-15 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Functional Mitral Regurgitation; Heart Failure
Keywords: Percutaneous mitral valve repair; Coronary sinus annuloplasty; Mitral loop cerclage
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single (Experimental): Intervention: Device: Mitral Loop Cerclage Annuloplasty with CSTV Protective Device
  Interventions: Device: Mitral Loop Cerclage Annuloplasty

INTERVENTIONS:
Device: Mitral Loop Cerclage Annuloplasty
  Other Names: MLC series (MLC-B-45-75-R and other 11 models)

SUMMARY:
To evaluate safety and feasibility of Mitral Loop Cerclage(MLC) Annuloplasty with CSTV for repair of functional mitral regurgitation.

DETAILED DESCRIPTION:
The objective of this prospective, single-center, open label, feasibility test is to assess the safety and efficacy of Mitral Loop Cerclage Annuloplasty with CSTV protective device in treating functional mitral regurgitation (FMR) associated with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* NYHA(New York Heart Association) Class III - IV, and symptomatic severe functional MR by 2014 ACC/AHA guideline in spite of optimal medical treatment.

(For optimal medical treatments, ①ACE inhibitor or angiotensin receptor blocker ②β-blocker ③ aldosterone antagonists should be given for at least 3 months unless the subject has contraindication for each drug)

Exclusion Criteria:

* Primary Mitral Regurgitation
* LV ejection fraction lower than 25%
* Creatinine ≥2.0 mg/dL
* Anomaly of Coronary Sinus
* Pre-existing devices in coronary sinus such as Implantable Cardioverter Defibrillator and Pacemaker
* 2:1 Atriventricular AV block or higher AV block and ventricular tachycardia
* Subjects with functional MR who need CABG or AVR performed
* Subjects who have functional MR caused by aortic valve disease
* Subjects who have uncontrollable hyperthyroidism
* Subjects who have severe TR due to primary valve leaflet disease
* Subjects who cannot be screened by cardiac CT
* Subjects who have possibility of coronary artery pinching even with Mitral Loop Cerclage system judged by cardiac CT
* Subjects who are unable to take anti-platelet agents
* Subjects who are participated in other clinical trials within 1 month of enrollment
* Subjects who have coagulation disorders
* Subjects who have thrombosis and embolism
* Subjects who are pregnant, or lactating, or plan pregnancy during the clinical trials
* Subjects who are deemed not to be eligible in this study by physician's discretion

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change of mitral regurgitation severity by regurgitant volume (RV) and effective regurgitant orifice (ERO) | 1 month
Change in mitral annulus geometry (septal lateral dimension) | 1 month
Rate of adverse events as a measure of safety | 1 month
  Rate of composite endpoint of MACE (Major Adverse Cardiac Event)
  * Death, myocardial infarction, cardiac tamponade, device related cardiac surgery, stroke

SECONDARY OUTCOMES:
Change of mitral regurgitation severity by regurgitant volume (RV) and effective regurgitant orifice (ERO) | 6 months
Change in mitral annulus geometry (septal lateral dimension) | 6 months
Change in mitral valve hemodynamics | 6 months
Change in left ventricle volumes | 6 months
Change in subjects' symptoms referred to NYHA (New York Heart Association) Classification System | 6 months
Technical success rate of the implantation and technical feasibility | 6 months
Rate of adverse events as a measure of safety | 6 months
  Rate of composite endpoint of MACE (Major Adverse Cardiac Event)
  * Death, myocardial infarction, cardiac tamponade, device related cardiac surgery, stroke

CONTACTS AND LOCATIONS:
Overall Officials: June-Hong Kim, MD, Ph D, Principal Investigator — Pusan National University Yangsan Hospital
Locations (2):
- National Institues of Health, Bethesda, Maryland, United States
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

REFERENCES:
- [Background] Kim JH, Kocaturk O, Ozturk C, Faranesh AZ, Sonmez M, Sampath S, Saikus CE, Kim AH, Raman VK, Derbyshire JA, Schenke WH, Wright VJ, Berry C, McVeigh ER, Lederman RJ. Mitral cerclage annuloplasty, a novel transcatheter treatment for secondary mitral valve regurgitation: initial results in swine. J Am Coll Cardiol. 2009 Aug 11;54(7):638-51. doi: 10.1016/j.jacc.2009.03.071. PMID 19660696
- [Result] Park YH, Chon MK, Lederman RJ, Sung SC, Je HG, Choo KS, Lee SH, Shin ES, Kim JS, Hwang KW, Lee SY, Chun KJ, Kim CM, Kim JH. Mitral Loop Cerclage Annuloplasty for Secondary Mitral Regurgitation: First Human Results. JACC Cardiovasc Interv. 2017 Mar 27;10(6):597-610. doi: 10.1016/j.jcin.2016.12.282. PMID 28335897